CLINICAL TRIAL: NCT02763332
Title: Effect of the Kinesio Taping in Patients With Fibromyalgia.
Brief Title: Effect of the Kinesio Taping in Fibromyalgia.
Acronym: EffKtFbm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Dr, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID012
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Efficacy; Taping
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Upper trunk group (UTG) (Experimental): In the UTG, the bandage was applied over the superior fibbers of the trapezious and levator scapulae muscle using a strip in a 'Y' shape. The individuals were asked to remain in an upright sitting position and the base of the strip was attached to the skin beyond the acromion without any tension. Later, we placed the two straps of the bandage with a range of tension from 15 to 25%. The main goal of this shape is achieve muscular relaxation of the trapezius, scapula levator and supraspinatus.
  Interventions: Other: Upper trunk group (UTG)
- Global trunk group (GTG) (Active Comparator): In the GTG the bandage was applied parallel to the paravertebral muscles in a 'C' shape. The individuals were sit in the same position with the head in the neutral position. The strip was pasted with approximately 25% of tension all over the paravertebral musculature. The main goal was procuring a global mechanical correction of the superior part of the trunk.
  Interventions: Other: Global trunk group (GTG)

INTERVENTIONS:
Other: Upper trunk group (UTG) — This bandage was placed over the upper trapezius muscle.
  Other Names: Upper trunk
  Arms: Upper trunk group (UTG)
Other: Global trunk group (GTG) — This bandage was placed globally along the back
  Other Names: Global trunk
  Arms: Global trunk group (GTG)

SUMMARY:
The prevalence of the fibromyalgia is about 10-15% in the European countries. It is unclear the etiology and pathogenesis of the syndrome. Several factors such as dysfunction of the central and autonomic nervous systems, neurotransmitters, hormones, immune system, external stressors, psychiatric aspects, and others seem to be involved. But the symptom commonly expressed by the people who suffer from it is pain.

The main goal of the present study is to analyse the effect of the kinesiotaping on the pain, comfort and postural position of the patient with fibromyalgia.

DETAILED DESCRIPTION:
All of the participants were recruited, in a non-probabilistic way, from the Valencian Association of Affected of Fibromyalgia from date to april 2016. Inclusion criteria include: age between 18 and 70 years old and diagnosis of fibromyalgia based on the American College of Rheumatology (ACR) diagnostic criteria. Once they expressed their interest in taking part of the study, potential participants underwent an examination by a rheumatologist of the association to confirm the diagnosis of fibromyalgia. People with other different diagnosis, musculoskeletal or neurological disorders that prevented the follow-up study, infections, whiplash, migraine, skin hypersensitivity or heart devices were excluded.

The participants were randomly allocated (random numbers table) to two different groups depending on the placement of the Kinesio Tape © (KT) by a physiotherapist which did not participated in the study. Thus, one group was composed by 18 women and was called "Upper trunk group" (UTG). The other group, composed by 17 women and called "Global trunk group" (GTG).

Patients were informed about the purpose of the study, procedures and risks, and they provided written informed consent before the treatment. The study protocol was approved by the authors´ University Ethic Committee where the study was conducted. All procedures were conducted in accordance to the Declaration of Helsinki.

A prospective, randomized, double blind, controlled trial was carried out. Participants were assessed two times, one before the intervention and another afterwards. They received a treatment of kinesiotaping during three weeks. Participants came to our laboratory each week in order to change their bandage and assure the adherence to the treatment.

The physiotherapist who conducted the assessments was blinded to the treatment received by the patients and the statistician was completely blinded to the goals of the study. The physiotherapist who applied the treatment had an extensive experience Kinesio Tape ©.

All enrolled participants were aware that they could receive two types of treatments but did not know the purposes of each treatment. They were instructed to not change their daily routines.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years old and diagnosis of fibromyalgia based on the American College of Rheumatology (ACR) diagnostic criteria (Wolfe et al., 2011). Once they expressed their interest in taking part of the study, potential participants underwent an examination by a rheumatologist of the association to confirm the diagnosis of fibromyalgia.

Exclusion Criteria:

* People with other different diagnosis, musculoskeletal or neurological disorders that prevented the follow-up study, infections, whiplash, migraine, skin hypersensitivity or heart devices were excluded.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity | three weeks
  The pain intensity was recorded by a visual analogue scale (VAS) of pain. The pain was expressed on a scale of 0-10, with 0 being "no pain" and 10 "maximum tolerable pain."

SECONDARY OUTCOMES:
Comfort. | three weeks
  Five VAS were used to identify their level of comfort in the following corporal regions: head-neck, shoulders, thoracic segment, lumbar region and pelvic region (0=absolute discomfort and 10=full comfort). Participants placed a mark along the line in order to measure their comfort level, which was scored to the nearest centimeter.
Impact on quality of life. | three weeks
  The Fibromyalgia Impact Questionnaire (FIQ) was used to assess the functional status of this population. This questionnaire is composed of 10 questions. Items 4 through 10 are horizontal linear scales marked in 10 increments on which the patient rates work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety and depression.
Physical well-being | three weeks
  Was determined using self-administered questionnaire, designed for this purpose included a 16-item. The reliability of the questionnaire was analyzed by Cronbach's alpha coefficient, which indicated a good internal consistency (α = 0.70).
Trunk posture. | three weeks
  To assess the position of the superior part of the trunk, the evaluation of the minor pectoral length in supine position was employed, taking the distance (with a tape measure) between the posterior edge of the acromion to the stretcher while the patients remain in that position with their hands laying on their belly.
Perception of change | three weeks
  Was evaluated with the Patient's Global Impression of Change scale after treatment. Participants were asked to score their perception of changing after the intervention received with a one-item questionnaire with seven alternatives (1= maximum change to 7 = no change at all).

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Espí-López, PhD, Principal Investigator — Faculty of Physiotherapy
Locations (1):
- Faculty of Physiotherapy, Valencia, Valencia, Spain

REFERENCES:
- [Result] Lim EC, Tay MG. Kinesio taping in musculoskeletal pain and disability that lasts for more than 4 weeks: is it time to peel off the tape and throw it out with the sweat? A systematic review with meta-analysis focused on pain and also methods of tape application. Br J Sports Med. 2015 Dec;49(24):1558-66. doi: 10.1136/bjsports-2014-094151. Epub 2015 Jan 16. PMID 25595290
- [Result] Mostafavifar M, Wertz J, Borchers J. A systematic review of the effectiveness of kinesio taping for musculoskeletal injury. Phys Sportsmed. 2012 Nov;40(4):33-40. doi: 10.3810/psm.2012.11.1986. PMID 23306413